CLINICAL TRIAL: NCT03214796
Title: Effect of Albumin Infusion on Oxidative Albumin Modification, Albumin Binding Capacity and Plasma Thiol Status
Acronym: ALB-INFUS
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: ALB-INFUS
Record Dates: First submitted 2017-06-12; First posted 2017-07-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Serum Albumin, Human; Albumins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, neutrophil granulocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Albumin infusion: Patients with decompensated cirrhosis and an indication for routine human albumin infusion
  Interventions: Drug: Human albumin

INTERVENTIONS:
Drug: Human albumin — Infusion of human albumin
  Other Names: Albumin

SUMMARY:
The aim of this study is to investigate the effect of albumin infusion on oxidative albumin modification, on plasma thiol status and on albumin binding capacity for DS in patients who routinely receive albumin infusion for various indications and to relate these findings with neurohumoral parameters, bacterial products such as endotoxin, and neutrophil function

DETAILED DESCRIPTION:
Albumin infusion has been shown to improve outcome in spontaneous bacterial peritonitis, to reverse hepatorenal syndrome combined with vasoconstrictors, and to prevent post-paracentesis circulatory dysfunction. These beneficial effects are associated with hemodynamic improvement reflected by neurohumoral changes such as a decrease in plasma renin activity .

Albumin is a multifunctional protein. Its biological functions include maintenance of oncotic pressure, solubilization and transport of hydrophobic substances, antioxidant function via its free sulfhydryl group at cysteine-34, metal binding at its N-terminus, immunomodulation and/or endothelial stabilization via binding and inactivation of endotoxin. Thus the beneficial effects of albumin infusion described above are probably not only due to plasma volume expansion but also to an improvement of various aspects of albumin function.

Albumin harbours two specific binding sites described by Sudlow: site I which binds large heterocyclic compounds and dicarboxylic acids (such as bilirubin) and site II which binds aromatic carboxylic compounds (such as benzodiazepines). Decreased binding of dansylsarcosine (DS) - a model ligand for the benzodiazepin binding site II - was found in patients with end-stage liver disease. Interestingly, extracorporeal albumin dialysis using the molecular adsorbents recirculating system (MARS) has been found to improve DS binding, while no such data exist for albumin infusion under the above-mentioned conditions.

Further examples for impaired albumin function in cirrhosis include alterations in fatty acid binding (as estimated by electron paramagnetic resonance) and impaired metal binding (measured as ischemia-modified albumin).

Impaired albumin function may be caused by oxidative albumin damage, which has been found in several disease conditions including chronic liver failure. Three fractions of albumin can be discerned according to the redox state of cysteine-34: non-oxidized human mercaptalbumin (HMA) with Cys-34 as free sulfhydryl, reversibly oxidized human nonmercaptalbumin-1 (HNA1) with Cys-34 as mixed disulfide, and irreversibly oxidized human nonmercaptalbumin-2 (HNA2) with Cys-34 oxidized to sulfenic, sulfinic or sulfonic acid. The investigators of this study have previously reported marked oxidative albumin damage in decompensated cirrhosis and even more so in acute-on-chronic liver failure and these alterations were found to be related to prognosis.

Small thiol compounds such as cysteine/cystin or glutathion interacting with the sulfhydryl group at Cys-34 may change the oxidation state of albumin and may be oxidized/reduced themselves. The role of small thiol compounds in various disease conditions and their putative alterations following albumin infusion is currently unknown. Due to the complex logistics of blood sample handling plasma thiol status is measured in a subset of 10 patients only.

While free Cys-34 of albumin accounts for about 80% of the antioxidant capacity of human plasma, both reversible and irreversible oxidation at this site will markedly reduce the antioxidant function of albumin. Besides, irreversibly oxidized albumin causes intense modifications of albumin structure and leads to marked alterations of albumin binding function.

Interestingly, oxidative albumin modification observed in chronic liver failure was paralleled by an impairment of albumin binding capacity as measured by DS binding. This finding among others has led to the concept of effective albumin concentration, which may further aggravate hypoalbuminemia observed in chronic liver failure.

The effect of albumin infusion on oxidative albumin modification and albumin function in chronic liver failure is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Routine indication for albumin infusion
* Informed consent

Exclusion Criteria:

* Malignant ascites
* Presence of hepatocellular carcinoma or advanced extrahepatic neoplasia
* Nephrotic syndrome
* Pregnancy, lactation
* Albumin infusion >80g within the last 48 hours

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Forty consecutive patients receiving albumin infusions routinely in the above-mentioned clinical conditions (paracentesis, hepatorenal syndrome, SBP) will be studied at the Medical University of Graz.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Albumin oxidation status | 48 hours
  changes in albumin oxidation status (HMA, HNA1, HNA2; percentage) due to albumin infusion measured by HPLC

SECONDARY OUTCOMES:
albumin binding capacity for dansylsarcosine | 48 hours
  changes in albumin binding capacity (IC50) due to albumin infusion
Plasma renin activity | 48 h
  changes in plasma renin activity (ELISA; uU/ml) due to albumin infusion
Plasma copeptin concentration | 48 h
  changes in plasma copeptin concentration (ELISA; pmol/l) due to albumin infusion
Plasma thiol status | 48 h
  changes in plasma thiol status (HPLC, umol/l) due to albumin infusion
serum endotoxin levels | 48 h
  changes in serum endotoxin levels (measured by HEK blue LPS detection kit, IU/ml) due to albumin infusion
Neutrophil phagocytic capacity | 48 h
  changes in neutrophil phagocytic capacity (flow cytometry; percentage FITC positive cells) due to albumin infusion
Neutrophil oxidative burst | 48 h
  changes in neutrophil oxidative burst (flow cytometry; percentage FITC positive cells) due to albumin infusion

CONTACTS AND LOCATIONS:
Overall Officials: Rudofl E Stauber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided